CLINICAL TRIAL: NCT01036061
Title: A Placebo-controlled, Single Blind, Randomized Two Part Study Toinvestigate the Tolerability, Pharmacokinetics, and brainDopamine D3 Receptor Occupancy of Increasing Repeat Doses ofGSK618334 for up to 21 Days in Healthy Volunteers.
Brief Title: GSK618334 Repeat Dose Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: 108414
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Substance Dependence
Keywords: compulsive discorders; addiction
MeSH Terms: conditions — Substance-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- GSK618334 low Dose (Experimental): GSK618334 Low Dose
  Interventions: Drug: GSK618334 Low Dose; Drug: GSK618334 PET subjects
- GSK618334 Medium Dose (Experimental): GSK618334 medium dose arm
  Interventions: Drug: GSK618334 PET subjects; Drug: GSK618334 Medium Dose
- GSK618334 High Dose (Experimental): GSK618334 High Dose Arm
  Interventions: Drug: GSK618334 PET subjects; Drug: GSK618334 High Dose
- GSK618334 Placebo (Experimental): Placebo for all 3 dose levels
  Interventions: Drug: GSK618334 Low Dose; Drug: GSK618334 Medium Dose; Drug: GSK618334 High Dose

INTERVENTIONS:
Drug: GSK618334 Low Dose — GSK618334 low dose
  Arms: GSK618334 Placebo; GSK618334 low Dose
Drug: GSK618334 PET subjects — PET subjects
  Arms: GSK618334 High Dose; GSK618334 Medium Dose; GSK618334 low Dose
Drug: GSK618334 Medium Dose — Medium Dose
  Arms: GSK618334 Medium Dose; GSK618334 Placebo
Drug: GSK618334 High Dose — GSK618334 High Dose
  Arms: GSK618334 High Dose; GSK618334 Placebo

SUMMARY:
The proposed study will evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics of repeated oral doses of GSK618334 in healthy male and female volunteers.

DETAILED DESCRIPTION:
GSK618334 strongly binds to dopamine type 3 receptors in the human brain and is being developed as an innovative treatment for substance dependence. This study will evaluate the safety, tolerability, blood concentrations and effect following repeated oral doses of GSK618334 in healthy male and female volunteers. The effect of food on a single oral dose of GSK618334 will also be evaluated. Another portion of this study will investigate dopamine type 3 receptor binding in the human brain by PET scan before and after repeated doses of GSK618334.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Males and Females between the ages of 18-50 years old
* Male and Female subjects must agree to use protocol specified contraceptive methods.
* Male subjects only in PET parts of the study.
* Capable of providing written informed consent.

Exclusion Criteria:

* A positive test for Hepatitis B or Hepatitis C within 3 months of screening.
* Current or chronic history of liver disease, or known liver/bile/gallbladder abnormalities.
* Personal or family history of heart disease (such as irregular heart beats, a history of sudden unexplained death in a first degree relative, or unexplained fainting).
* Screening ECG parameters outside the protocol specified parameters.
* Pulse rate <50 or >100 bpm OR a systolic blood pressure >140 or <95 mmHg OR a diastolic blood pressure >90 or <50 mmHg at screening and/or baseline.
* Pregnant or lactating females.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Previous inclusion in a research and/or medical protocol involving nuclear medicine, PET or radiological investigations with significant radiation burden.
* Significant suicidal risk.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2009-09-28 (Actual); Primary Completion 2010-02-17 (Actual); Study Completion 2010-02-17 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability endpoints will be: adverse events, laboratory values, cardiovascular variables (blood pressure, heart rate, ECG), temperature, respiratory rate, assessment of mood and abnormal movements, and GSK618334 blood levels. | First dose to follow-up
To assess blood concentrations of GSK618334 after repeated oral doses. | First dose to 72 hours post last dose

SECONDARY OUTCOMES:
To assess the effect of food on GSK618334 blood concentrations after a single dose. | First dose of the single dose session to 24 hours after dosing of the repeat dose session
The dopamine type 3 receptor binding in the brain (by PET scan) of GSK618334 following the repeat dose session. | First dose to 24 hours after last dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 108414 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/108414?search=study&search_terms=108414#rs
- Available data/document: Statistical Analysis Plan: 108414 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 108414 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 108414 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 108414 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 108414 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 108414 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register